CLINICAL TRIAL: NCT02267694
Title: A Trial of Freeze-dried Black Raspberry in Maintenance of Remission of Ulcerative Colitis
Brief Title: Study of Freeze-dried Black Raspberry in Maintenance of Ulcerative Colitis
Acronym: BRB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRB113728
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Black raspberry powder (Other): Black raspberry powder 25 grams once daily for 4 weeks. If tolerated, will increase to 25 grams twice a day for another 20 weeks. Total length of active treatment 24 weeks.
  Interventions: Drug: Freeze-dried black raspberry powder

INTERVENTIONS:
Drug: Freeze-dried black raspberry powder

SUMMARY:
This research study is about adding Black Raspberry powder to the treatment regimen of patients with ulcerative colitis who are currently in remission and doing well.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years of age) with known diagnosis of ulcerative colitis who are currently in remission on a stable dose of 5-ASA products and/or steroids (equivalent to prednisone 20 mg or less). English speaking/reading male or female patients from all ethnicities will be considered for the study.

Exclusion Criteria:

* Treatment with Immunomodulators and/or biologic agents, active disease flare, patients younger than 18 years old, patients who are pregnant or trying to get pregnant, breast feeding and those with reported history of allergy or hypersensitivity to berry products.

Patients who are using NSAIDS will also be excluded from the study but low dose ASA (81-162 mg) is permitted if needed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10-05 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
Remission rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Haleh Vaziri, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States